CLINICAL TRIAL: NCT03647215
Title: A Cohort Study To Establish the Prevalence of Mutations in Patients With CML Who Meet the ELN Criteria for Warning or Failure and Patients With Ph+ ALL With Detectable BCR-ABL Currently Being Treated With First or Subsequent TKI Therapy in the UK, Ireland, or France Using Next-Generation Sequencing
Brief Title: CALLS: CML and Ph+ALL Low Level Mutation Prevalence Survey
Status: Completed | Type: Observational
Sponsor: Incyte Biosciences UK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Other Study IDs: INCB 84344-401
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia; Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Keywords: Chronic myeloid leukemia; chronic phase; accelerated phase; blast phase; Philadelphia chromosome-positive acute lymphoblastic leukemia; tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with CML and Ph+ALL who are being treated with their first or subsequent TKI therapy. CML patients must meet the ELN criteria for warning and failure ) or have high SOKAL score (>0.8) or presence of additional chromosomal abnormalities (ACAs) and have detectable BCR-ABL levels. Ph+ALL patients need detectable BCR-ABL levels only.

SUMMARY:
A multicenter, prospective cohort study of the mutation status of patients with chronic myeloid leukemia (CML) and Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) who are being treated with first or subsequent tyrosine kinase inhibitor (TKI) therapy in the UK, Ireland, or France.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) with CML (in all phases of disease) or Ph+ ALL with detectable BCR-ABL levels who are being treated with a first or subsequent TKI.
* Patients with CML must meet the warning or failure criteria as per the ELN guidelines for first second and subsequent treatment line, including:

  * BCR-ABL/ABL IS transcripts > 10% at 3 months
  * BCR-ABL/ABL IS transcripts > 1% at 6 months
  * BCR-ABL/ABL IS transcripts > 0.1% at 12 months or later
* Patients with CML must not currently be in MMR (ie, have disease with BCR-ABL1/ABL1 transcripts > 0.1% IS).

OR

* Patients with Ph+ ALL with any level of BCR-ABL/ABL IS transcripts. Patients with Ph+ ALL should have BCR-ABL1/ABL1 transcript levels > 0.1% and should not be currently enrolled in UKALL14 but may have relapsed during or after participation in UKALL14.
* Patients with an intermediate or high Sokal score (> 0.8) can be recruited into the study from 3 months after diagnosis, irrespective of BCR-ABL1/ABL1 transcript levels at 3 months.
* Patients with additional chromosomal abnormalities at diagnosis and patients with AP-CML may be recruited into the study, irrespective of BCR-ABL1/ABL1 transcript levels at 3 months and beyond provided BCR-ABL1/ABL1 transcript levels are > 0.1% IS. It is recommended that these patients have mutational analysis performed every 3 months irrespective of BCR-ABL1/ABL1 transcript levels until they reach MR3/MMR (BCR-ABL1/ABL1 < 0.1% IS).
* Any patients who have previously undergone testing for KD mutations, irrespective of KD mutational analysis test results.
* Patients who have the ability to understand the requirements of the study and provide written informed consent.

Exclusion Criteria:

Patients without detectable BCR-ABL and patients who have switched TKI due to intolerance but who have met the criteria for optimal response (CP-CML, ELN 2013 guidelines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 50 centers in the UK, Ireland and France that treat adult patients with CML and Ph+ ALL will be selected for participation in the study. The sites selected will be a mixture of hospital and academic centers.
  The target study population will include adult patients with CML who meet the ELN criteria for warning or failure or have high SOKAL score > 0.8 or presence of additional chromosomal abnormalities (ACAs), all with detectable BCR-ABL levels. Ph+ ALL patients must have detectable BCR-ABL levels. Patients will be taking their first or subsequent TKI.
  Consecutive patients within each prescriber's practice who meet the enrollment criteria and provide informed consent will be invited to enroll into the study.
  Repeat NGS KD mutation testing is permitted under the protocol as deemed part of the standard management of patients.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with any mutation | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.
Frequency of all specific mutations | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.

SECONDARY OUTCOMES:
Percentage of participants with individual mutations in chronic phase (CP)-CML, accelerated phase (AP)-CML, and blast phase (BP)-CML | Up to approximately 1 month per individual participant.
  Participants in all phases of CML (CP, AP, and BP) will be enrolled.
Frequency of individual mutations in chronic phase (CP)-CML, accelerated phase (AP)-CML, and blast phase (BP)-CML | Up to approximately 1 month per individual participant.
  Participants in all phases of CML (CP, AP, and BP) will be enrolled.
Percentage of participants with individual mutations in Ph+ ALL | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.
Frequency of individual mutations in Ph+ ALL | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.
Percentage of participants with individual mutations by whether a participant is intolerant or resistant to their previous TKI | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.
Frequency of individual mutations by whether a patient is intolerant or resistant to their previous TKI | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS.
Percentage of participants with individual mutations by BCR-ABL level | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS. BCR-ABL levels defined as > 0.1% to 1% international scale (IS), > 1% to 10% IS, > 10% IS.
Frequency of individual mutations by BCR-ABL level | Up to approximately 1 month per individual participant.
  All samples will be processed by NGS. BCR-ABL levels defined as > 0.1% to 1% international scale (IS), > 1% to 10% IS, > 10% IS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thompson, MD, Study Director — Incyte Biosciences UK
Locations (33):
- Ireland (2):
  - Limerick University Hospital, Limerick, Dooradoyle
  - University Hospital Waterford, Waterford
- United Kingdom (31):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Derriford Hospital, Plymouth, Devon
  - Broomfield Hospital Chelmsford, Chelmsford, Essex
  - Queen's Hospital, Romford, Essex
  - Aberdeen Royal Infirmary, Aberdeen, Foresterhill
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Medway Maritime Hospital, Gillingham, Kent
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Royal Oldham Hospital, Manchester, Lancashire
  - Queens Medical Centre, Nottingham, Nottinghamshire
  - Ipswich Hospital, Ipswich, Suffolk
  - Heart of England NHS Foundation Trust, Birmingham, West Midlands
  - Russells Hall Hospital, Dudley, West Midlands
  - St Bartholomew's Hospital, London, West Smithfield
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire
  - Monklands Hospital, Airdrie
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital Wales, Cardiff
  - Croydon University Hospital, Croydon Health Services NHS Trust, Croydon
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy's Hospital, London
  - King's College Hospital, London
  - The James Cook University Hospital, South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS FT, Sheffield
  - Royal Stoke University Hospital, Cancer Centre, University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Undecided
Blood samples will be identifiable by a code consisting of numbers and initials. Samples may be stored and tested for up to 5 years after the completion of the study.